CLINICAL TRIAL: NCT00613535
Title: Magnetic Resonance Imaging and Clinical Outcomes After Three Different Treatments for Articular Cartilage Lesions Concomitant With Partial Meniscectomy
Brief Title: Knee Articular Cartilage Debridement in Conjunction With Partial Meniscectomy
Acronym: MILE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The correlation coefficient at the interim analysis with results for all three groups pooled, did not reach the level of statistical significance of (p<0.05).
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-706-DHH; 1093528
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Torn Meniscus
Keywords: Partial Meniscectomy; Partial Thickness Knee Tear; MR Imaging; Mechanical Debridement; Crepitus; Stability; Coblation; Bipolar Radiofrequency; Debridement; Recurrent Knee Pain; meniscectomy; meniscus; cartilage lesion; articular cartilage lesion; articular cartilage; knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lavage debridement to remove loose fragments (Active Comparator): Articular cartilage defect left untreated by surgical tool during partial meniscectomy
  Interventions: Procedure: Lavage debridement
- Mechanical Debridement (Active Comparator): Remove large chondral flaps and loose fragments
  Interventions: Device: Mechanical debridement
- RF based Debridement (Active Comparator): Debridement to remove loose fragments followed by use of Paragon T-2 RF wand to smooth the base of the shoulder of the tear
  Interventions: Device: Paragon T2; Device: RF- based Debridement

INTERVENTIONS:
Device: Mechanical debridement — Mechanical shaver will be used to remove large chondral flaps and loose fragments
  Arms: Mechanical Debridement
Device: Paragon T2 — Use Paragon device to debride after removal of larger chondral lesion flaps with mechanical shaver.
  Arms: RF based Debridement
Procedure: Lavage debridement — Remove loose chondral fragments
  Arms: Lavage debridement to remove loose fragments
Device: Mechanical Debridement — Use of a mechanical device such as a shaver, punch, or biter to remove large chondral flaps and loose fragments
  Arms: Mechanical Debridement
Device: RF- based Debridement — Use of debridement device to remove large fragments followed by use of RF-based debridement to smooth the base of the shoulder of the tear.
  Arms: RF based Debridement

SUMMARY:
The aim of this study is to describe changes at the site of the study patient's articular cartilage lesion on the femoral condyle with multiple magnetic resonance imaging (MRI) outcomes 6 months after treatment using one of three standard surgical treatment methods: 1) lavage debridement; 2) mechanical debridement; 3) mechanical and radiofrequency-based debridement.

DETAILED DESCRIPTION:
Fibrillated articular cartilage are commonly detected during arthroscopy when treating knee pathologies such as a torn meniscus or a damaged anterior cruciate ligament (ACL). The severity of these lesions is graded using a scheme such as the International Cartilage Research Society (ICRS) classification system. Grade I lesions are often left untreated, while Grade IV lesions require dedicated surgical intervention. Grade II and III lesions are frequently treated when they are encountered arthroscopically.

Currently, it is not known whether treatment of fibrillated articular cartilage is beneficial or whether one procedure is superior to another. Magnetic resonance imaging is the best technique currently available for non-invasive assessment of chondral lesions. The primary aim of the proposed study is to compare post-procedure MR imaging characteristics of fibrillated articular cartilage treated using one of the three standard of care measures: 1) Washing of the knee joint with saline solution to clear blood, fluid or loose tissue (also known as lavage); 2) Lavage in addition to mechanical shaver (a manual surgical tool used by the study doctor); and 3)Lavage in addition to the Paragon device (RF-based microdebridement), which may also be used with a mechanical (or manual) surgical tool. The secondary aim is to determine the association between imaging features and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:Screening

* Age between 18 and 60 years
* BMI <35
* Meniscal tear (medial or lateral) diagnosed by H+P exam and/or imaging in the index knee
* No severe joint space narrowing (IKDC Classification) seen on weight-bearing AP X-ray in the index knee
* No avascular necrosis in the index knee as evidenced by preop MRI obtained within 6 months prior to randomization
* No Varus (>10 degrees) or Valgus (>15 degrees)knee deformities as seen by AP X-ray in the index knee
* Minimal or no abnormality of contralateral knee as shown by clinical exam and/or imaging
* Candidate for unilateral arthroscopic treatment of the knee
* Visual Analog Scale (VAS) pain score of 30 mm or greater in the index knee at the time of screening
* Must be able to undergo MRI at required time points per appendix D
* Physically and mentally willing and able to comply with study requirements
* Must be willing and able to follow the standardized rehabilitation protocol (Appendix C)
* Subject must sign IRB approved informed consent form

Arthroscopy Inclusion Criteria:

* Arthroscopic confirmation of ICRS Grade II or III chondral lesion on the medial or lateral femoral condyle

Exclusion Criteria: Screening

* Knee instability, malalignment, or patellar tracking dysfunction in the index knee
* Inflammatory rheumatoid arthritis or other systemic inflammatory arthritis in the index knee or contralateral knee
* Previous total meniscectomy in the index knee
* Previous surgical treatment of the index knee by arthroscopy less than 2 years prior to treatment by this study
* Previous total meniscectomy
* Previous knee tendon and/or ligament repair or patellar surgery of index knee
* Previous microfracture or bone marrow stimulation of the index knee
* Previous unsuccessful osteotomy in the index knee
* Presence of fractures, osteocysts or osteolysis in the index knee
* Presence of osteoarthritis in the index knee
* Pre-existent osteoarthritis of weight-bearing joints (e.g. hips or contralateral knee) that adversely affects gait
* Participation in another clinical study
* Terminally ill
* Drug therapy for the index knee with systemic steroid therapy, steroid intra-articular therapy or intra-articular hyaluronic acid therapy within 2 months of enrollment into this study
* Receiving narcotic pain medication by prescription for other conditions unrelated to knee injury
* Contralateral knee involvement causing abnormal ambulation and non-compliance with rehabilitation
* Pregnant or suspected pregnant
* Coagulation disorder or patient is receiving anti-coagulants, which cannot be safely stopped for 14 days (7 days prior to surgery and 7 days post-surgery)

Arthroscopy Exclusion Criteria:

* Presence of Grade IV chondromalacia anywhere in the index knee
* ACL, PCL or MCL tear of the index knee
* Osteochondritis dissecans (OCD)of the index knee
* Meniscal tear requiring total meniscectomy
* Evidence of osteoarthritis in the index knee

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
In vivo magnetic resonance imaging (MRI) features of the femoral condyle chondral lesion | 6 months after arthroscopy

SECONDARY OUTCOMES:
To determine whether recovery from recurrent pain, effusion, localized mechanical symptoms, and quality of life are equivalent for treatment groups | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Pettrone, M.D., Principal Investigator — Commonwealth Orthopaedics
Locations (10):
- United States (10):
  - HOPE Research Institute, Phoenix, Arizona
  - Kerlan Jobe Orthopaedic Foundation, Los Angeles, California
  - JDP Medical Research, Aurora, Colorado
  - Colorado Orthopedic Consultants, P.C., Englewood, Colorado
  - Shrock Orthopedic Research, LLC, Fort Lauderdale, Florida
  - University of Mass. Memorial Medical Center, Worcester, Massachusetts
  - University of Rochester Medical Center Department of Musculoskeletal Research, Rochester, New York
  - Basin Orthopedic Surgical Specialists, Odessa, Texas
  - Commonwealth Orthopaedics, Arlington, Virginia
  - Anderson Clinic, Arlington, Virginia

REFERENCES:
- [Background] Figueroa D, Calvo R, Vaisman A, Carrasco MA, Moraga C, Delgado I. Knee chondral lesions: incidence and correlation between arthroscopic and magnetic resonance findings. Arthroscopy. 2007 Mar;23(3):312-5. doi: 10.1016/j.arthro.2006.11.015. PMID 17349476
- [Background] Hjelle K, Solheim E, Strand T, Muri R, Brittberg M. Articular cartilage defects in 1,000 knee arthroscopies. Arthroscopy. 2002 Sep;18(7):730-4. doi: 10.1053/jars.2002.32839. PMID 12209430
- [Background] Widuchowski W, Widuchowski J, Trzaska T. Articular cartilage defects: study of 25,124 knee arthroscopies. Knee. 2007 Jun;14(3):177-82. doi: 10.1016/j.knee.2007.02.001. Epub 2007 Apr 10. PMID 17428666
- [Background] Sgaglione NA, Miniaci A, Gillogly SD, Carter TR. Update on advanced surgical techniques in the treatment of traumatic focal articular cartilage lesions in the knee. Arthroscopy. 2002 Feb;18(2 Suppl 1):9-32. doi: 10.1053/jars.2002.31783. PMID 11828343
- [Background] Brittberg M, Winalski CS. Evaluation of cartilage injuries and repair. J Bone Joint Surg Am. 2003;85-A Suppl 2:58-69. doi: 10.2106/00004623-200300002-00008. No abstract available. PMID 12721346
- [Background] Shelbourne KD, Jari S, Gray T. Outcome of untreated traumatic articular cartilage defects of the knee: a natural history study. J Bone Joint Surg Am. 2003;85-A Suppl 2:8-16. doi: 10.2106/00004623-200300002-00002. PMID 12721340
- [Background] Alford JW, Cole BJ. Cartilage restoration, part 1: basic science, historical perspective, patient evaluation, and treatment options. Am J Sports Med. 2005 Feb;33(2):295-306. doi: 10.1177/0363546504273510. PMID 15701618
- [Background] Messner K, Maletius W. The long-term prognosis for severe damage to weight-bearing cartilage in the knee: a 14-year clinical and radiographic follow-up in 28 young athletes. Acta Orthop Scand. 1996 Apr;67(2):165-8. doi: 10.3109/17453679608994664. PMID 8623573
- [Background] Fowler P. Arthroscopic lavage or debridement did not reduce pain more than placebo did in patients with osteoarthritis. J Bone Joint Surg Am. 2003 Feb;85(2):387. doi: 10.2106/00004623-200302000-00038. No abstract available. PMID 12571328
- [Background] Owens BD, Stickles BJ, Balikian P, Busconi BD. Prospective analysis of radiofrequency versus mechanical debridement of isolated patellar chondral lesions. Arthroscopy. 2002 Feb;18(2):151-5. doi: 10.1053/jars.2002.29906. PMID 11830808
- [Background] Barber FA, Iwasko NG. Treatment of grade III femoral chondral lesions: mechanical chondroplasty versus monopolar radiofrequency probe. Arthroscopy. 2006 Dec;22(12):1312-7. doi: 10.1016/j.arthro.2006.06.008. PMID 17157730
- [Background] Mithoefer K, Williams RJ 3rd, Warren RF, Potter HG, Spock CR, Jones EC, Wickiewicz TL, Marx RG. The microfracture technique for the treatment of articular cartilage lesions in the knee. A prospective cohort study. J Bone Joint Surg Am. 2005 Sep;87(9):1911-20. doi: 10.2106/JBJS.D.02846. PMID 16140804
- [Background] Henderson IJ, Tuy B, Connell D, Oakes B, Hettwer WH. Prospective clinical study of autologous chondrocyte implantation and correlation with MRI at three and 12 months. J Bone Joint Surg Br. 2003 Sep;85(7):1060-6. doi: 10.1302/0301-620x.85b7.13782. PMID 14516048
- [Background] Voloshin I, Morse KR, Allred CD, Bissell SA, Maloney MD, DeHaven KE. Arthroscopic evaluation of radiofrequency chondroplasty of the knee. Am J Sports Med. 2007 Oct;35(10):1702-7. doi: 10.1177/0363546507304328. Epub 2007 Jul 20. PMID 17644661
- [Background] Yetkinler DN, Greenleaf JE, Sherman OH. Histologic analysis of radiofrequency energy chondroplasty. Clin Sports Med. 2002 Oct;21(4):649-61, viii. doi: 10.1016/s0278-5919(02)00015-7. PMID 12489295